CLINICAL TRIAL: NCT04368676
Title: Breath Regulation and Yogic Exercise An Online Therapy for Calm and Happiness (BREATH): an RCT for Frontline Hospital and Long-term Care Home Staff Managing the COVID-19 Pandemic
Brief Title: Breath Regulation and Yogic Exercise An Online Therapy for Calm and Happiness During the COVID-19 Pandemic
Acronym: BREATH
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Art of Living Foundation (Unknown)
Responsible Party: Principal Investigator, Akshya Vasudev, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 115855
Record Dates: First submitted 2020-04-26; First posted 2020-04-30 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Job Stress; Workplace Stress; Compassion Fatigue; Psychological Trauma; Healthcare Workers; Healthcare Providers
Keywords: COVID-19; Coronavirus; Healthcare staff; Work stress; insomnia; anxiety; depression; resilience; mind-body intervention
MeSH Terms: conditions — Occupational Stress; Compassion Fatigue; Psychological Trauma; COVID-19; Coronavirus Infections; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will be blinded to the treatment hypothesis while the data analyst will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sudarshan Kroya Yoga (SKY) (Experimental): Sudarshan Kriya Yoga (SKY) will be delivered using the Hospital approved Cisco WebEx platform. The online version of SKY will be delivered by at least one certified Canadian SKY teacher, with at least one back up teacher, under the supervision of Ms. Ronnie Newman, Director of Research and Health Promotion, Art of Living Foundation, USA. The online version of SKY for healthcare workers has a total duration of 10.5 hours. This includes 3 interactive online sessions of 2.5 hours each during the first week followed by four weekly follow-up sessions each 30-45 minutes long. For ease of scheduling, multiple time windows will be offered.
  Interventions: Other: Sudarshan Kriya Yoga (SKY)
- Health Enhancement Program (HEP) (Active Comparator): The Health Enhancement Program (HEP) will be delivered using the Hospital approved Cisco WebEx platform. The online version of HEP for healthcare workers has a total duration of 10.5 hours. This includes 3 interactive online sessions of 2.5 hours each during the first week followed by four weekly follow-up sessions each 30-45 minutes long. For ease of scheduling, multiple time windows will be offered. HEP will be taught by Dr. Paris Lai, co-investigator and senior psychiatry resident.
  Interventions: Other: Health Enhancement Program

INTERVENTIONS:
Other: Sudarshan Kriya Yoga (SKY) — The SKY program is a standardized, easy to learn sequential breathing yoga consisting of regulated breathing techniques followed by a timed rhythmic breathing practice. Participants will learn various exercises including rhythmic breathing, gentle yoga, and guided meditation.
  Arms: Sudarshan Kroya Yoga (SKY)
Other: Health Enhancement Program — HEP is a structured group program designed to help participants with information and instruction how to lead a healthier life. Participants will be provided psychoeducation and support regarding healthy active living using techniques like music therapy, diet control, exercise, and monitoring these via journaling.
  Arms: Health Enhancement Program (HEP)

SUMMARY:
This study will examine the feasibility of conducting an online Randomized Controlled Trial (RCT) in frontline hospital and long term care healthcare staff in managing COVID-19 patients in London, ON. The study will randomize participants to Sudarshan Kriya Yoga (SKY) or a Health Enhancement Program (HEP).

DETAILED DESCRIPTION:
The COVID-19 pandemic continues to escalate as a global health threat, leading to devastating impacts on the healthcare system. Frontline healthcare workers are dealing with increased demands and fears for their own, as well as their family's safety. Adding to the stress is the limited ability to maintain social connectedness as physical distancing measures are in place. The investigators plan to conduct an open-label feasibility randomized controlled trial (RCT), comparing an online breath based yogic intervention called Sudarshan Kriya Yoga (SKY) (n=30) versus an online control mind-body intervention called the Health Enhancement Program (HEP) (n=30) in 60 hospital and long term care frontline staff that are managing COVID-19 patients. Participants will be blinded to the treatment hypothesis while data analyst will be blinded to treatment allocation. Both SKY and HEP will be taught online in two phases in the first week followed by weekly reinforcement sessions for the following 4 weeks. Feasibility measures will be assessed as well as self-rated measures of insomnia, anxiety, depression, and resilience. The investigators expect that it will be feasible to conduct an online RCT of two mind-body interventions, SKY and HEP, in staff managing the COVID-19 pandemic, and that the investigators will be able to remotely monitor safety and efficacy of these interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be frontline hospital or long-term care home staff involved in the management of COVID-19 patients in Canada or The United States of America.
2. Participants will be aged 18 to 70.
3. Participants will be willing and able to attend, via WebEx software, the introductory phase of SKY or HEP, as well as at least two of the four weekly follow-up sessions
4. Have sufficient hearing to follow verbal instructions.
5. Have an adequate understanding of English.
6. Able to sit without physical discomfort for 60 minutes.
7. Not pregnant and willing to remain not pregnant for the duration of the study.

Exclusion Criteria:

1. Inability to independently provide informed consent.
2. Current suicidality as assessed by the suicide item of the Patient Health Questionnaire-9 scale.
3. History of bipolar disorder.
4. History of chronic PTSD.
5. History of schizophrenia or schizoaffective disorder.
6. Currently practice any type of formal meditation, mindfulness, or breathing techniques regularly (greater than 3 times per week).
7. History of complex PTSD.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
Rate of participant recruitment | 1 year
  The number of participants recruited per month will be calculated as a feasibility measure.
Rate of retention | 1 year
  The retention rate of participants will be calculated as a feasibility measure.
Completeness of data entry | 1 year
  The completeness of study assessments will be assessed as a feasibility measure by calculating the missing percentage of data in case report forms.
Cost of interventions | 1 year
  The cost of both study interventions will be calculated to assess the total study cost for interventions and the cost per participant. This information will be used as a feasibility measure.
Unexpected costs | 1 year
  The total of unexpected costs will be calculated as a feasibility measure.

SECONDARY OUTCOMES:
Change in Athens Insomnia Scale | Change from Week 0 to week 3 and to week 5
  The Athens Insomnia Scale will be used to assess insomnia. This scale is an 8-item, self-rated measure of the extent of sleep difficulties over the last 30 days with each item representing a different aspect of sleep (e.g. "Overall Quality of Sleep"). Ratings are from 0 to 4, with 0 being no difficulty with the item and 4 being the most difficulty with the item. Higher overall scores on this scale indicate higher difficulties with sleep.
Change in Generalized Anxiety Disorder 7-item scale | Change from Week 0 to week 3 and to week 5
  The Generalized Anxiety Disorder 7-item scale (each scored 0-3) is a self-rated measure of anxiety and has been validated for the diagnosis of Generalized Anxiety Disorder in the adult population. Scores range from 0 to 21. Higher scores indicate greater anxiety symptoms (5-9, mild anxiety; 10-14, moderate anxiety; 15-21 severe anxiety).
Change in Patient Health Questionnaire 9 | Change from Week 0 to week 3 and to week 5
  The Patient Health Questionnaire (PHQ-9) is a 9-item, self-rated measure of depression which has been validated for screening a major depressive episode in adults. Total scores indicate various levels of depression: 0-4, no depression; 5-9, mild depression; 10-14, moderate depression; 15-19, moderately severe depression; 20-27, severe depression.
Change in Connor-Davidson Resilience Scale | Change from Week 0 to week 3 and to week 5
  The Connor-Davidson Resilience Scale (CD-RISC) is a brief self-rated assessment tool that comprises of 10 items, each rated on a 5-point Likert scale (0 = not true at all to 4 = true nearly all the time). Higher scores reflect greater resilience, which is a measure of one's ability to cope with stress. The scale demonstrated strong reliability and validity and has been studied in a variety of populations including medical personnel, nurses, social workers and physicians).

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai KSP, Watt C, Ionson E, Baruss I, Forchuk C, Sukhera J, Burhan AM, Vasudev A. Breath Regulation and yogic Exercise An online Therapy for calm and Happiness (BREATH) for frontline hospital and long-term care home staff managing the COVID-19 pandemic: A structured summary of a study protocol for a feasibility study for a randomised controlled trial. Trials. 2020 Jul 14;21(1):648. doi: 10.1186/s13063-020-04583-w. PMID 32665041
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860